CLINICAL TRIAL: NCT03408821
Title: Examining the Feasibility and Effectiveness of Case Manager Delivered Problem Solving Therapy on Late Life Depression: An Open-label Prospective Pilot Study
Brief Title: CM Delivered PST in LLD Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Bell Let's Talk Community Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4698
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Late Life Depression

STUDY DESIGN:
Intervention Model Description: Participants will attend 8 weekly sessions of Case Manager delivered Problem Solving Therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problem Solving Therapy (Experimental): All participants will attend 8 weekly sessions of Case Manager delivered Problem Solving Therapy.
  Interventions: Other: Problem Solving Therapy (PST)

INTERVENTIONS:
Other: Problem Solving Therapy (PST) — Participants will attend 8 weekly session of Case Manager (CM) implemented PST, a form of group talk therapy.

SUMMARY:
This study seeks to determine the feasibility and efficacy of a Problem Solving Therapy intervention for the treatment of late life depression (LLD). Participants diagnosed with LLD will participate in 8 weekly sessions of Problem Solving Therapy, a form of talk-therapy, over a period of eight weeks. A Case Manager (CM) trained in this therapy will lead the PST sessions. Participants will attend a clinical assessment pre and post study intervention to assess depression severity, quality of life, anxiety, insomnia, functional disability, and participant's acceptability of the intervention. Additionally self-rated depression will be collected weekly over 8 weeks.

DETAILED DESCRIPTION:
The study will be a single-centre, open-label, longitudinal, pragmatic, pilot trial. Research participants at this site will be 40 men and women between the ages of 60 and 85 who have mild to moderate major depressive disorder (MDD). Participants will be recruited from primary, secondary and tertiary care centres in London, Ontario and surrounding areas. Study participation will involve 10 study visits over a total of 10 weeks. This includes 8 weekly sessions of case manager (CM) implemented Problem Solving Therapy (PST) over a period of 8 weeks and 2 clinical assessment visits pre and post intervention.

PROBLEM-SOLVING THERAPY INTERVENTION: PST is a minimally invasive treatment. This intervention will be taught in groups of approximately 10 individuals. The eight sessions of CM implemented PST will involve psychotherapy also known as talk therapy between the CM's and study participants in a group setting. Psychogeriatric interdisciplinary staff (CM's) i.e. psychiatric nurses, social workers, occupational therapists, and recreation specialists who have been previously trained in PST will function in the roles of facilitator, cofacilitator and scribe. The roles can be shared amongst the professionals to build capacity in each role or maintained over time if so desired. Sessions will be approximately one-and-a-half to two hours in length and conducted at libraries in London, ON. The first meeting will be informal in which the staff and potential group participants will be welcomed, introductions made, group rules regarding confidentiality discussed, an overview of problem solving approach described and the depression/problem solving cycle introduced. Participants will be told of the relationship between effective problem solving and changes in feelings of depression and anxiety. At the second meeting group participants will be welcomed to the initial problem solving session, group rules of confidentiality reviewed again and then each of the participants will be asked to describe important psychosocial aspects of their lives in the previous week. Facilitation will be kept to a minimum with questions designed to encourage further exploration of problems experienced. The staff person acting as the scribe shall make notes of each participant's comments. Once all the group members have checked in, the scribe shall summarize problems that have been mentioned. One of the participants will be then asked to volunteer to act as the problem solver over the next week and if there is a particular problem that they are interested in completing. Once a volunteer has identified the problem it will be listed on a flipchart and the group shall take a ten minute break. After the break, the problem will be discussed again to ensure that the correct problem has been determined. Then the goal shall be listed on the flipchart and solutions to the problem will be discussed. Once they are listed the group shall review each and note the reasons why this is a good choice and the reasons why this may not be a good choice. Considerations include effort required, time commitment, emotional impact, the need to involve others and desirability from the participants perspective. Then the participant shall narrow the options and make a decision about what solutions he/she will try in the next week. An action plan will be then developed to achieve the solutions e.g. what is the first step, when will it be made, any resources that are needed before beginning the problem solving. In addition, the participant will be asked to engage in pleasant activities on a daily basis noting the date, activity and rate how satisfied the activity made them feel on a scale of 0 to 10 with 0= Not at all and 10=Super. At the third meeting, the facilitator shall ask the participant who volunteered to solve a problem to report to the group first. That person would have made notes about their experience and use these as a reference to report back to the group. Some may make diagrams to describe their experience and share these with the group. Each session shall continue using the above format and participants will be encouraged to volunteer at least one time to practice the problem solving approach. As the group continues to meet, there will be more peer support evident as the participants begin to know each other, realize their common bonds and experience a sense of community within the group setting. The final meeting will be a time to celebrate the accomplishments of the group, listing all of the problems mentioned and those solved by the participants and an opportunity to share social time together. Participants will be asked to complete a Patient Health Questionnaire (PHQ-9) at the beginning of the initial problem solving session and continue to do so at each session. The facilitator shall comment on the changes in the scores and shall ask the participants if their experience mirrors the scores, their anxiety and depression or not. Each time point will provide an opportunity to remind the group of the depression - problem solving cycle. The CM's will teach the participant's a structured approach to cope with and resolve issues in the participant's life. Using the six stages of problem resolution including: a) identifying and clarifying the problem b) setting clear achievable goals c) brain-storming to generate solutions d) selecting a preferred solution e) clarifying steps to implement solutions, and f) evaluation. Focus will be on issues the study participant currently has in their life and not on problems from their past.

SCREENING AND INITIAL ASSESSMENTS: Potential participants will be provided a Letter of Information (LOI) and given at least 24 hours to review the letter. The Research Assistant (RA) will then contact potential participants by phone and pre-screen these participants for potential eligibility using the Patient Health Questionnaire-2 (PHQ-2). This is essential so that participants who will not be eligible do not unnecessarily travel to the hospital for screening. Those participants who score a 0 on the PHQ-2 will not be invited to a screening assessment. The screening assessment will begin with a review of the LOI, an opportunity for the potential participant to ask any questions, and a signing of the LOI by both the participant and a witness. Participants will then be screened as per inclusion and exclusion criteria by the RA, administered a Mini Mental State Exam, section A of a Mini-International Neuropsychiatric Interview (MINI), and a Hamilton Depression Rating Scale (HAM-D17). Participants meeting eligibility criteria at this point will be invited to participate in this study. This initial assessment shall also include administration of a Cumulative Illness Rating Scale for Geriatrics (CIRS-G), EuroQol 5 Dimension 5 level (EQ-5D-5L), Athena Insomnia Scale, World Health Organization Disability Assessment Schedule 2 (WHODAS-2), and a Generalized Anxiety Disorder (GAD-7). Following the final PST session participants will be asked to return for a final assessment with the RA. This post intervention assessment will include a HAM-D17, EQ-5D-5L, Athens Insomnia Scale, WHODAS-2, a GAD-7, and a likert scale to measure acceptability. At each PST session the CM's will ask participant's to complete a Patient Health Questionnaire-9 (PHQ-9) to assess changes in depressive symptoms. These questionnaires will be provided to the RA by the CM's following completion of the group's intervention, so that this data can be included in the studies final report. Following the first groups and last groups completion a focus group will be conducted. This focus group will collect qualitative data to determine long-term sustainability of PST for seniors in London, ON and surrounding area. The focus group will be lead by a research staff member who has experience with focus group interviews and qualitative study design.

ELIGIBILITY:
Inclusion Criteria:

Participants will be considered eligible for the study if they:

1. Are of either gender and 60 years of age or greater.
2. Reside in a community setting (either independent living environment or retirement home).
3. Meet diagnostic criteria for major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) criteria.
4. Have a Hamilton Depression Rating Scale (HAMD) 17-item total score of >= 8 and < 24 at baseline.
5. Have a Mini Mental Status Exam score of >= 25.
6. Have adequate hearing and vision to be able to participate in Problem Solving Therapy, with no significant sensory impairment
7. Fluent in English both written and oral.

Exclusion Criteria:

Participants will be considered ineligible for participating in the study if they:

1. Have suicidal ideation requiring inpatient admission to hospital for stabilization.
2. Have an unstable medical condition requiring hospital admission.
3. Have a life expectancy of less than 6 months or are currently receiving palliative care.
4. Have psychotic symptoms.
5. Have a lifetime history of bipolar disorder or schizophrenia.
6. Are currently alcohol dependent or have another substance dependence.
7. Are diagnosed with moderate to severe dementia.
8. Are planning admission to a long-term care facility within next 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Successful implementation of Problem Solving Therapy (PST). | 10 weeks
  The primary outcome measure will be if CM delivered PST can be successfully implemented in the London Health Sciences Centre geriatric outreach program. If the recruitment goal of n=40 is met within 1 year, and 60% of participants complete the PST program, missing no more than 3 of the 8 weekly follow-ups, the primary objective will be considered to be met.

SECONDARY OUTCOMES:
Depression severity as measured by the Hamilton Depression Scale (HAM-D17) | Week 0, week 9.
  The HAM-D17 rates symptoms commonly associated with Major Depressive Disorder (MDD). A total score is calculated based on the first 17 questions of the HAM-D with a score range of 0 to 53. A higher score indicates more severe depression, and a lower score indicates fewer and/or less severe symptoms of depression. This assessment will be completed pre and post study intervention.
Quality of life as measured by the EuroQol 5 Dimension 5 level (EQ-5D-5L). | week 0, week 9.
  The European Quality of Life (EQ-5D-5L) scale will be used to assess the quality of life of study participants. This scale has two scores; the descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system consists of 5 questions each with 5 possible answers allowing for 5 possible health states. A score of 1 indicates no problems with the 5 measured dimensions, while a score of 5 would indicate the most severe possible state for each dimension. The descriptive system includes 5 sub-scores ranging from 1 (no issues) to 5 (severe problems), which will be converted to a specific single index value. The EQ VAS consists of only one question ranging from 0 (worst possible state of health) to 100 (best possible state of health).This assessment will be completed pre and post study intervention.
Anxiety severity as measured by the Generalized Anxiety Disorder 7-item (GAD-7) scale. | week 0, week 9.
  The GAD-7 rates anxiety severity based on 7 questions with scores ranging from 0 to 21. A higher score indicates more severe anxiety, and a lower score indicates less sever anxiety.This assessment will be completed pre and post study intervention.
Insomnia severity as measured by the Athens Insomnia Scale. | week 0, week 9.
  The Athens Insomnia scale measures sleep difficulty over the previous month with scores ranging from 0 to 24. A higher score indicates more severe insomnia while a lower score indicates less difficulty sleeping. This assessment will be completed pre and post study intervention.
Functional disability as measured by the World Health Organization Disability Assessment Schedule 2 (WHODAS-2). | week 0, week 9.
  The WHODAS-2 is a 36 item questionnaire used to assess disability that covers 6 domains of functioning; cognition, mobility, self-care, getting along, life activities, and participation. Scores range from 0 to 100 and are reported as a percentage, with higher scores indicating more disability and lower scores indicating less disability. This assessment will be completed pre and post study intervention.
Depression Severity as measured by the Patient Health Questionnaire-9 (PHQ-9). | 8 weeks
  The PHQ-9 contains 9 questions that rate the severity of depression. Scores range from 0 to 27 with more severe scores indicating a higher severity of depression. This assessment will be completed weekly by participants during each study intervention session.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There are no plans in place at this time to share individual participant data.